CLINICAL TRIAL: NCT06184620
Title: Correlation Between Angle Closure Glaucoma Data and Lens Zonule Status
Status: Completed | Type: Observational
Sponsor: Guangfu Dang (Other)
Responsible Party: Sponsor-Investigator, Guangfu Dang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(047)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Primary Angle Closure Glaucoma
Keywords: primary angle closure glaucoma; UBM; lens zonule
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PACG group: All patients in the experimental group met the diagnostic criteria of primary angle-closure glaucoma in the Chinese Glaucoma Guidelines(2020).
- control group: The depth of the anterior chamber is normal, and the whole corner of the chamber is open; The cup-to-plate ratio is less than 0.5; No family history of glaucoma

SUMMARY:
The goal of this observational study is to discuss the correlation between primary angle-closure glaucoma and the state of the suspended ligament of the lens and the pathogenesis of PACG by measuring the biological data of primary angle-closure glaucoma and observing its anatomical changes.

DETAILED DESCRIPTION:
Patients clinically diagnosed with Primary angle-closure glaucoma (PACG) and normal control patients from December 2020 to January 2022 were enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* The depth of the anterior chamber is normal, and the whole corner of the chamber is open;
* The cup-to-plate ratio is less than 0.5;
* No family history of glaucoma.

Exclusion Criteria:

* Previous history of trauma or internal eye surgery in both eyes or one eye;
* Used "pilocarpine", "atropine" and other drugs to change the size of the pupil and the shape of the chamber Angle within 1 week;
* Combined with other eye diseases affecting the Angle and suspension ligament, such as uveitis, ciliary cyst, high myopia, retinal diseases, etc.;
* Can not cooperate with UBM and Angle scopy;
* Refuse to participate in this researcher.

Ages: 47 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From December 2020 to January 2022, patients with primary angle-closure glaucoma and normal control patients were diagnosed for the first time and intended to undergo cataract surgery in the ophthalmology department of the First Affiliated Hospital of Shandong First Medical University (Shandong Qiandfo Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Axial Length (AL), Lens Thickness (LT),Lens Vault (LV), Pupil Diameter (PD), | before operation
  Axial Length (AL), Lens Thickness (LT),Lens Vault (LV), Pupil Diameter (PD),
Anterior Chamber Depth (ACD) in seat and rectum position, White To White (WTW), pupil vault (LV), pupil diameter (PD), The Lens Zonular Length (LZL) and Angle Opening Distance at 500μm (AOD500) in the upper, lower, nasal and temporal directions | before operation
  Anterior Chamber Depth (ACD) in seat and rectum position, White To White (WTW), pupil vault (LV), pupil diameter (PD), The Lens Zonular Length (LZL) and Angle Opening Distance at 500μm (AOD500) in the upper, lower, nasal and temporal directions

CONTACTS AND LOCATIONS:
Locations (1):
- guangfu Dang, Jinan, Shandong, China